CLINICAL TRIAL: NCT05671666
Title: Ureagenesis Analysis in Healthy Subjects and in Urea Cycle Disorder Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ureagenesis01352
Record Dates: First submitted 2022-11-01; First posted 2023-01-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-03

CONDITIONS: Urea Cycle Disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy controls or UCD patients (Other)
  Interventions: Diagnostic Test: Urea cycle flux study

INTERVENTIONS:
Diagnostic Test: Urea cycle flux study — Quantification of ureagenesis

SUMMARY:
Urea cycle disorders (UCDs) are dramatic congenital inherited metabolic disorders. There is no cure. Many novel therapeutic approaches are currently being developed, which hopefully will change the current situation. Testing the efficacy of such new therapies in patients is a challenge, because many clinical parameters are influenced by several disturbances and biochemical parameters are often not very specific.

The measurement of ureagenesis is a tool to analyze the entire function of the urea cycle in a single test. This is more meaningful for the characterization of UCD patients than the analysis of single metabolites or enzymes. Therefore, the test will be important to evaluate current and future novel therapies.

The term "ureagenesis" means "production of urea", which is the main task of the urea cycle. This total urea production can be measured with a "tracer" (in this case a stable ammonium chloride isotope). This tracer is non-radioactive and non-toxic. It is for example used as an unmarked substance in cough syrup, diuretic drugs and as food additive. Thus, the tracer does not pose a risk to the participant, especially since only a very low dose is applied.

The investigators will analyze specific substances from the urea cycle (namely [15N, 14N] urea and several [15N] amino acids) that are produced during the test and compare them with results from healthy people. Venous and capillary blood will be sampled at 15 to 30 minutes intervals up to 2 hours after administration of the stable isotope tracer. The maximum test duration is 5 hours.

This project is being carried out at one site, namely the University Children's Hospital in Zurich.

This project is being carried out under Swiss law. The responsible Ethics Committee has reviewed and approved the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects at any age and given written informed consent
* subjects with a UCD confirmed by genetic or enzymatic diagnostics at any age and given written informed consent

Exclusion Criteria:

* healthy subjects with acute and chronic disease requiring treatment of any kind
* pregnant or lactating women.
* UCD patients with acute and chronic (other than her/his UCD) disease requiring treatment
* UCD patients in which intake of carglumic acid cannot be stopped for 24 hours prior to the test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of flux through the urea cycle using stable isotopes in healthy subjects and patients, and the change of rate of flux through the urea cycle in patients after an intervention or for follow-up. | Baseline for healthy subjects and patients and post-intervention (up to 1 year after the intervention) for patients
  Measurement of total concentrations of urea in plasma (in mmol/L) and amino acids in plasma (in micromol/L) and their enrichment (in %) after application of a stable isotope tracer by using a high-resolution liquid chromatography mass spectrometry (LC MS) method.

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No